CLINICAL TRIAL: NCT06777407
Title: Brief Mindfulness-Based Intervention to Reduce Psychological Distress in Health Sciences Students At a Public University in Peru
Brief Title: Brief Mindfulness-Based Intervention to Reduce Psychological Distress in Health Sciences Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of San Marcos, Peru (Other)
Responsible Party: Principal Investigator, Leonardo Rojas Mezarina, Telehealth Unit Coordinator, National University of San Marcos, Peru
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0222-2023
Record Dates: First submitted 2024-10-19; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-09

CONDITIONS: Mindfulness; Psychological Distress
Keywords: Health Sciences Students; Mindfulness; Psychological Distress

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Information on self-care and managing psychological distress, along with 8 weeks of synchronous virtual sessions (1.5 hours per week), will be provided as part of the brief mindfulness-based intervention.
  Interventions: Behavioral: Brief Mindfulness-Based Intervention to Reduce Psychological Distress
- Control group (Other): Information on self-care and managing psychological distress will be provided to help participants develop strategies for coping with mental health challenges effectively.
  Interventions: Other: Psychoeducational brochure

INTERVENTIONS:
Behavioral: Brief Mindfulness-Based Intervention to Reduce Psychological Distress — The brief mindfulness-based intervention is an eight-week training program designed for groups of 15 to 20 participants. The weekly sessions will last 90 minutes for the first session and 60 minutes for the following seven sessions. The program will be led by a certified mindfulness trainer, who is not part of the research team and will be solely responsible for training-related activities.
  Arms: Intervention Group
Other: Psychoeducational brochure — Information on self-care and managing psychological distress will be provided. Once the study is completed and the data has been collected, participants in the control group will receive the intervention.
  Arms: Control group

SUMMARY:
This project aims to evaluate the effectiveness of a brief mindfulness-based intervention in reducing psychological distress among first-year health sciences students at the Universidad Nacional Mayor de San Marcos. The study will be a randomized controlled trial, comparing the effects of the intervention on psychological distress and mindfulness with standard treatment. Additionally, it will assess the acceptability of the virtual intervention, considering current limitations and the growing importance of digital tools.

DETAILED DESCRIPTION:
General Objective To evaluate the effectiveness of a brief mindfulness-based intervention in reducing psychological distress in first-year health sciences students at UNMSM.

Hypothesis The average psychological distress score of first-year health sciences students at UNMSM who receive the mindfulness-based intervention will be lower compared to those who do not receive it.

The average mindfulness score of first-year health sciences students at UNMSM who receive the intervention will be higher compared to those who do not receive it.

Unit of Analysis First-year health sciences students from the Faculty of Medicine at UNMSM during the 2023 academic year.

Sampling The sampling will be non-probabilistic and convenience-based, including all students who wish to participate in the study.

Sample Size The sample size will consist of 60 participants per group, calculated using the formula for comparing two repeated means in two distinct groups.

Procedures

Participant Recruitment

Recruitment will take place during the month prior to the start of the intervention through invitations sent to institutional emails, the Faculty of Medicine's social media, text messages to students' cell phones (with prior authorization), and announcements in general classes. Participants will be enrolled during a one-week registration period, where they will complete an informed consent form and an initial assessment, which will include the following questionnaires:

Sociodemographic data sheet Perceived Stress Scale (PSS-13) Depression Symptoms Scale (PHQ-9) Mindfulness Scale (MAAS-5) Randomization

Participants will be randomly assigned to two groups using a random number generator:

Intervention Group (A): Will receive the brief mindfulness-based intervention, consisting of eight synchronous virtual sessions of 60 minutes once per week, along with a psychoeducational brochure.

Control Group (B): Will only receive the psychoeducational brochure and will be offered the intervention after the ninth week, once the study is completed.

Intervention

Content: The intervention is a mindfulness training program conducted in groups of 15 to 20 participants over eight weeks. The first session will be 90 minutes long, while the remaining sessions will last 60 minutes.

Program Implementation: A certified mindfulness trainer, not part of the research team, will guide the sessions. The program will be conducted over a two-month period with a total of 120 participants.

Evaluations Assessments will be conducted at the start of the intervention (M1) and at the end of the eight weeks (M2) using self-administered questionnaires. The primary outcome will be the scores on the Perceived Stress Scale, and secondary outcomes will include the Depression Scale, the Mindfulness Scale, and the Acceptability Scale (only in M2).

Analysis Plan

Primary Outcome: The treatment effect will be evaluated using a one-way ANOVA model, considering the variable defining the experimental and control group assignment as the treatment. Additionally, an analysis of covariance (ANCOVA) will be applied to account for the baseline outcome value as a covariate and adjust for potential residual confounding variables despite randomization. Effect sizes (η² and partial η²) will be calculated within the same model with 95% confidence intervals. Since a cluster effect may exist within the intervention subgroups, the intraclass correlation coefficient will be calculated to determine whether a multilevel model is necessary to adjust variance due to the cluster effect.

Secondary Outcome: A comparison of means between the experimental and control groups will be conducted.

Other Details: In the event of participant loss, results will be shown using an intention-to-treat analysis and compared with results analyzed according to protocol. All analyses will be conducted using R 4.2 (CRAN R Project).

ELIGIBILITY:
Inclusion Criteria:

Undergraduate health sciences students (from the schools of medicine, nursing, midwifery, nutrition, and medical technology) in their first year.

Students who have completed the initial pre-intervention assessment. Students who have signed the informed consent form. Students aged 18 years or older.

Exclusion Criteria:

Students with a score greater than 20 on the PHQ-9 scale (indicating severe depressive symptoms) at the time of the pre-intervention assessment.

Students with any other severe mental illness or a high risk of suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Psychological Stress | At the beginning of the study
  Psychological stress is an adaptive emotional response to threatening situations that enables individuals to respond effectively according to the environment or context. However, when this response becomes disproportionate in intensity, quality, or frequency, it can lead to discomfort and avoidance behaviors, negatively impacting a person's performance.
  The Escala de Percepción Global al Estrés (EPGE - 13) is a stress level measurement scale with two dimensions (one positive and the other negative) that has been adapted from previous versions with a greater number of items to this shorter 13-item scale that has been validated in different languages and different settings. In our environment it has been recently validated in university students resulting in an estimated reliability in the scores generated of a Cronbach's alpha of 0.79 for the eustress factor and 0.77 for the distress factor.

SECONDARY OUTCOMES:
Mindfulness | At the beginning of the study
  This innate ability has been shown to help individuals cope more effectively with stressful situations.
  The Mindful Awareness Attention Scale 5 (MAAS-5) is a brief adaptation of the original scale that has been validated in our environment with accepted levels of validity and reliability (omega coefficient 0.85) to measure mindfulness in university students. It consists of 5 items rated with Likert scale scores from 1 "almost always" to 6 "almost never", with higher scores indicating greater presence of the quality. The scale is in the public domain and does not require permission by the authors for its use for research purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universidad Nacional Mayor de San Marcos, Lima, Lima Province, Peru

IPD SHARING:
Plan to Share IPD: No